CLINICAL TRIAL: NCT06974539
Title: Optimization of PCaVision: A Prospective Study for CAD-based Detection of Clinically Significant Prostate Cancer Using mpUS and Contrast Agents
Brief Title: TULIP ReTrain Study
Acronym: TULIP ReTrain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Angiogenesis Analytics (Industry)
Responsible Party: Principal Investigator, Harrie P. Beerlage, Prof. Dr. H.P. Beerlage, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL-009343
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: mpUS; CEUS; PCaVision; CAD; Optison; Sonovue; radical prostatectomy; AI diagnosis
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiparametric ultrasound with contrast (Sonovue and Optison) (Other): Diagnostic test: Multiparametric ultrasound with contrast (Sonovue and Optison)
  Interventions: Diagnostic Test: Multiparametric ultrasound with contrast (Sonovue and Optison)

INTERVENTIONS:
Diagnostic Test: Multiparametric ultrasound with contrast (Sonovue and Optison) — Participants will receive 3D mpUS using both Sonovue and Optison contrast agents during a single transrectal imaging session.

SUMMARY:
This prospective clinical study aims to retrain and validate the PCaVision AI algorithm for the detection and localization of clinically significant prostate cancer (csPCa) using multiparametric ultrasound (mpUS) with two different ultrasound contrast agents: Sonovue and Optison. Data will be collected using a commercial version of the LOGIQ E10 ultrasound machine, with full histopathological correlation in patients undergoing radical prostatectomy.

DETAILED DESCRIPTION:
The PCaVision CAD system was initially developed using Sonovue contrast and a research-only ultrasound machine (LOGIQ E10 R3). In this study, the algorithm will be retrained using data acquired from the LOGIQ E10 R4, a commercially available system, and using both Sonovue and Optison as contrast agents. The goal is to enhance generalizability and enable broader clinical adoption. The study includes two cohorts: patients scheduled for radical prostatectomy (for training and voxel-level validation) and patients with a negative prostate MRI (for patient-level specificity evaluation). All participants will undergo 3D transrectal mpUS with both contrast agents in a single session. Full prostate histology from RP specimens will serve as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥18 years
* Cohort 1: Histologically confirmed prostate cancer scheduled for radical prostatectomy
* Cohort 2: Negative multiparametric prostate MRI (PI-RADS ≤ 2)

Exclusion Criteria:

* Severe pulmonary hypertension
* Cardiac right-to-left shunt
* Known allergy to Sonovue or Optison
* Contraindication for ultrasound contrast agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of PCaVision Algorithm (Sonovue and Optison) Compared to Histopathology | From baseline imaging to histopathology report (typically within 2-4 weeks post-surgery)
  Sensitivity and specificity of the PCaVision algorithm in detecting and localizing clinically significant prostate cancer (csPCa, Gleason Grade Group ≥2) at the voxel level, based on 3D multiparametric ultrasound (mpUS) images using Sonovue and Optison, validated against full prostate histology after radical prostatectomy.

SECONDARY OUTCOMES:
Specificity of PCaVision in MRI-Negative Cohort | From baseline imaging to completion of image processing and analysis (within 2 weeks of scan)
  Evaluation of the specificity of the PCaVision algorithm for csPCa detection at the patient level in men with a negative prostate MRI (PI-RADS ≤2), using mpUS imaging with Sonovue and Optison.
Diagnostic Performance Comparison Between Sonovue and Optison | Imaging and analysis completed within 4 weeks post-surgery
  Head-to-head comparison of diagnostic performance (sensitivity, specificity, AUC) of PCaVision on mpUS scans obtained with Sonovue versus Optison, using RP histopathology as reference. Evaluated at voxel level and using simulated biopsy protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Oddens, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared for this study because the imaging data and histopathology are linked to highly sensitive clinical records. Due to privacy concerns and the risk of re-identification, even in coded form, sharing of raw participant-level data is not planned. Data will only be used internally for algorithm development and validation under strict confidentiality agreements.

REFERENCES:
- [Background] Jager A, Zwart MJ, Postema AW, van den Kroonenberg DL, Zwart W, Beerlage HP, Oddens JR, Mischi M. Development and validation of a framework for registration of whole-mount radical prostatectomy histopathology with three-dimensional transrectal ultrasound. BMC Urol. 2025 Apr 3;25(1):73. doi: 10.1186/s12894-025-01736-4. PMID 40175990
- [Background] van den Kroonenberg DL, Jager A, Garrido-Utrilla A, Reitsma JB, Postema AW, Beerlage HP, Oddens JR. Clinical Validation of Multiparametric Ultrasound for Detecting Clinically Significant Prostate Cancer Using Computer-Aided Diagnosis: A Direct Comparison with the Magnetic Resonance Imaging Pathway. Eur Urol Open Sci. 2024 Jul 1;66:60-66. doi: 10.1016/j.euros.2024.06.012. eCollection 2024 Aug. PMID 39050912
- [Background] van Moorselaar RJ, Voest EE. Angiogenesis in prostate cancer: its role in disease progression and possible therapeutic approaches. Mol Cell Endocrinol. 2002 Nov 29;197(1-2):239-50. doi: 10.1016/s0303-7207(02)00262-9. PMID 12431818
- [Background] Jager A, Vilanova JC, Michi M, Wijkstra H, Oddens JR. The challenge of prostate biopsy guidance in the era of mpMRI detected lesion: ultrasound-guided versus in-bore biopsy. Br J Radiol. 2022 Mar 1;95(1131):20210363. doi: 10.1259/bjr.20210363. Epub 2021 Jul 29. PMID 34324383
- See also: Angiogenesis Analytics - cooperation partner — https://angiogenesisanalytics.com/